CLINICAL TRIAL: NCT03878329
Title: Randomized Prospective Trial of Telemedicine Based Remote Home Monitoring After Liver Transplantation
Brief Title: Telemedicine Based Remote Home Monitoring After Liver Transplantation
Acronym: TelehealthOLT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Shimul Shah, Professor of Surgery, Chief, Solid Organ Transplantation, Department of Surgery, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TelehealthOLT
Record Dates: First submitted 2019-03-14; First posted 2019-03-18 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Liver Failure; Liver Transplant; Complications
MeSH Terms: conditions — Liver Failure

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Masking Description: Non-blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard of care (No Intervention): standard of care treatment
- remote home monitoring (Experimental): use of telemedicine based remote home monitoring
  Interventions: Behavioral: remote home monitoring

INTERVENTIONS:
Behavioral: remote home monitoring — Will use telemedicine to guide behavior changes in outcomes
  Arms: remote home monitoring

SUMMARY:
A significant opportunity exists to involve patients and their caregivers in more effective perioperative care and transition to home for transplant patients. Stakeholders were engaged through the University of Cincinnati Liver Transplant Program to prioritize changes in improving post transplant care. The initial findings indicated that increasing "care between visits" is the top priority for patients for improving function, quality of life and independence. Building on existing telehealth research, an enhanced home management program (HMP) to leverage and improve patient self-care following liver transplantation was developed, specifically by improving adherence, reducing readmissions and improving the transition from hospital to home. The improvement of care may have profound effect in the first 90 days after transplant on important long-term health parameters that affect clinical outcomes such as depression, weight gain, blood pressure control and diabetes management. With patient engagement, a randomized controlled trial is proposed comparing traditional provider-based care vs. traditional care with HMP. These two arms will need 50 patients in each arm with a 0.5 year follow up. Patients have said that the primary outcomes are quality of life, function and independence. To that end, the primary study outcomes are assessment of adherence, readmissions (90-day), patient satisfaction. The HMP model will advise providers, health care systems, and transplant centers how to improve patient care, especially among those at greatest risk of poor outcomes specifically minorities and those of low socioeconomic status.

DETAILED DESCRIPTION:
The successful care of patients undergoing liver transplantation and support of their caregivers consumes significant personal, institutional and community resources before and after surgery. Depression and anxiety are common after transplant, leading to apprehension about the ability to care successfully for oneself and poor adherence with complex medication and health behavior regimens.1,2 Although a patient's quality of life improves immediately following transplantation, when compared with the general population the vast majority of liver transplant recipients have significant deficiencies in most quality of life domains.3,4 This is most evident in minorities and patients of low socioeconomic status who have difficulty adjusting to the demands of complex medical and surgical care and are challenged by lack of literacy and cultural bias.5-7 Indeed, the reoperation and readmission rate in the first 90 days are the highest of any surgery performed in the United States.8 Effective perioperative care is critical following surgery in this high acuity patient population. Optimizing care in the perioperative period should improve recovery and outcomes, including depression, general health maintenance and long-term adherence.9,10 While practice guidelines for care after liver transplant exist, they lack specifics and are based on outdated models that do not reflect patient preferences, needs or expectations. Improving current processes in health care delivery before and after liver transplantation is critical to optimize outcomes that matter: survival, function, and independence. The improvement of care may have profound effect in the first 90 days after transplant on important long-term health parameters that affect clinical outcomes such as depression, weight gain, blood pressure control and diabetes management.11 Through a stakeholder engagement process with the University of Cincinnati Liver Transplant Program designed to find ways to improve post transplant care, increasing "care between visits" is the top priority for patients to improve function, quality of life and independence. Patients said that medication adherence and hospital readmissions are their largest barrier to success, and that they believe care immediately post-transplant in the first 90 days is the most important determinant of long-term outcomes. A twenty-patient pilot program assessed the feasibility of a patient-designed telehealth monitoring program after liver transplant, and it met with an extraordinary level of enthusiasm by our patients. In this proposal, the ability of this home management program (HMP) will be tested, developed by patients for patients, to improve transition care from hospital to home and patient adherence with a self-care regimen following liver transplantation.

The medical community must develop innovative health delivery systems following complex surgeries like transplantation in order to maximize post-operative care, adherence to a new and complex self-care regimen, independence, and ultimately survival. Our proposed telehealth delivery model will optimize the quality, efficiency and outcomes of post-discharge care following liver transplantation. The HMP model will advise providers, health care systems, and transplant centers how to improve patient care, especially among those at greatest risk of poor outcomes, specifically minorities and those of low socioeconomic status. The objective of this proposal with the following specific aims:

Aim 1: Perform a randomized clinical trial to evaluate the impact of an enhanced, telehealth-based home management program (HMP) on medication and behavioral self-care adherence rates, and on 90-day and 1-year readmission rates following discharge for liver transplantation.

Hypothesis: Through enhanced patient engagement, HMP will increase medication and self-care adherence rates and reduce 90-day and 1-year readmission rates when compared to a traditional care model.

SubAim 1A: To determine whether underserved and minority patients achieve greater benefit from the HMP compared with more advantaged patient populations.

Aim 2: Evaluate the impact of the HMP on more distal clinical outcomes post liver transplantation including weight control, diabetes management, blood pressure regulation and depression.

Hypothesis: Enhanced home monitoring will have persisting health benefits beyond the 90-day time frame of the HMP intervention on a variety of chronic disease measures important in this population, including weight loss, diabetes management, blood pressure control, and depression.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects (≥ 18 years old) who are liver transplant recipients.
2. Discharged home within 45 days of liver transplant.
3. Able and willing to provide informed consent.

Exclusion Criteria:

1. Post-transplant admission and care provided by University of Cincinnati Medical Center or rehab facility > 45 days after liver transplant.
2. Unable to have 4G wireless connectivity or wifi in their home.
3. Patient has any form of psychiatric disorder or a condition that, in the opinion of the investigator, may hinder communication with the investigator.
4. Inability to cooperate or communicate with the investigator.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
90- day readmission | 90 days
  Assess readmission

IPD SHARING:
Plan to Share IPD: Yes
Protocol will be share
Supporting Information: Study Protocol
Time Frame: 1 year after study completed.
Access Criteria: investigator with HIPAA compliance

REFERENCES:
- [Result] Lee TC, Kaiser TE, Alloway R, Woodle ES, Edwards MJ, Shah SA. Telemedicine Based Remote Home Monitoring After Liver Transplantation: Results of a Randomized Prospective Trial. Ann Surg. 2019 Sep;270(3):564-572. doi: 10.1097/SLA.0000000000003425. PMID 31356267
- [Derived] Mellon L, Doyle F, Hickey A, Ward KD, de Freitas DG, McCormick PA, O'Connell O, Conlon P. Interventions for increasing immunosuppressant medication adherence in solid organ transplant recipients. Cochrane Database Syst Rev. 2022 Sep 12;9(9):CD012854. doi: 10.1002/14651858.CD012854.pub2. PMID 36094829